CLINICAL TRIAL: NCT05183087
Title: Pilot Study of Long-Term Effects of Repetitive, Low-Level Blast Exposure (RLLBE) on Special Operations Forces (SOF) Service Members
Brief Title: Long-Term Effects of Repetitive, Low-Level Blast Exposure on Special Operations Forces Service Members
Acronym: ReBlast
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Neurocritical Care Faculty and Associate Professor of Neurology, Massachusetts General Hospital
Other Study IDs: 2020P002695
Record Dates: First submitted 2021-12-09; First posted 2022-01-10 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Traumatic Brain Injury; Blast Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Blast Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Special Operations Forces (SOF) Personnel: n=30 SOF Personnel
  Interventions: Diagnostic Test: 3T Connectome MRI; Diagnostic Test: 7 Tesla MRI; Diagnostic Test: TSPO PET; Diagnostic Test: Tau PET; Diagnostic Test: Cognitive and Behavioral Assessments; Diagnostic Test: Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: 3T Connectome MRI — MRI scan of structural connectivity
Diagnostic Test: 7 Tesla MRI — MRI scan of functional connectivity
Diagnostic Test: TSPO PET — PET scan of neuroinflammation
Diagnostic Test: Tau PET — PET scan of tau deposition
Diagnostic Test: Cognitive and Behavioral Assessments — Assessments of memory, attention, complex reasoning, mood and other cognitive/behavioral domains
Diagnostic Test: Blood Biomarkers — Blood-based assessments of proteomic and metabolic biomarkers of brain injury

SUMMARY:
This is a pilot study to identify biomarkers that individually, and in combination, demonstrate the greatest sensitivity to repetitive, low-level blast exposure (RLLBE) neurotrauma in Special Operations Forces (SOF) personnel. The proposed cross-sectional, multimodal study will elucidate the potential effects of long-term RLLBE by comparing biomarkers across subjects.

DETAILED DESCRIPTION:
The proposal includes a comprehensive battery of assessments characterized by high-field neuroimaging, proteomics, and experimental cognitive and neurobehavioral evaluations, which will be implemented alongside standardized clinical diagnostic tools. The results will inform the design of a larger trial to validate the diagnostic utility of these biomarkers as well as their ability to predict RLLBE-related clinical outcomes. A secondary aim will be to define the underlying mechanisms, risk and resilience factors, and clinical phenotypes associated with RLLBE.

Biomarkers assessed over the course of a two-day evaluation will include:

1. 3 Tesla Connectome MRI to detect structural disruption of brain networks
2. 7 Tesla MRI to detect functional disruption of brain networks
3. Translocator protein (TSPO) PET - ligand [11C]-PBR28 to detect neuroinflammation
4. Tau PET - ligand [18F]-MK6240 to detect tau deposition
5. Neurocognitive assessments to detect signs of cognitive/behavioral dysfunction
6. Self-report indicators of cognitive/behavioral dysfunction
7. Blood biomarkers to detect evidence of blast injury using proteomics and metabolomics

We hypothesize that a multimodal assessment using Connectome MRI, 7 Tesla MRI, TSPO PET, Tau PET, cognitive/behavioral tests, proteomics and metabolomics will identify biomarkers of RLLBE-related brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 25-45 years of age
2. Males, regardless of race or ethnicity
3. Active duty Special Operation Forces
4. History of combat deployment confirmed by Veterans Affairs (VA) or Department of Defense (DOD) records (defined as: while serving in the U.S. military, individual was deployed to a region of conflict)
5. History of combat exposure during any deployment as measured by endorsement of any item on the Combat Exposure Scale (CES)

Exclusion Criteria:

1. History of moderate or severe traumatic brain injury (TBI) (using the VA/DOD definition: initial Glasgow Coma Scale score < 13, coma duration > ½ hr, post-traumatic amnesia duration > 24 hr, or abnormal structural brain imaging)
2. History of major neurologic disorder such as stroke or spinal cord injury resulting in a significant decrement in functional status or loss of independent living capacity
3. Untreated or unstable severe psychiatric condition (e.g., schizophrenia or bipolar disorder) that is likely to impact study participation or ability to complete study procedures
4. Current severe medical condition (excluding currently diagnosed mild TBI or concussion) that requires long-term treatments (e.g., cancer, diabetes mellitus, human immunodeficiency virus, autoimmune disorders)
5. Any cardiac, respiratory, or other medical condition that may affect cerebral metabolism
6. Benzodiazepines other than lorazepam, desmethyldiazepam and oxazepam within past month
7. MRI contraindications

   1. Metal in the body that would make an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye
   2. Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
   3. Inability to lie supine for up to 2 hours in the MRI scanner, as assessed by physical examination and medical history (e.g., back pain, arthritis)
   4. > 300 lbs (weight limit of the MRI table)
8. Prior radiation exposure of ≥ 50 mSv over the past 12 months, in the context of research, as determined by review of DOD medical records (e.g., prior imaging studies) and self-report
9. Any condition which, in the opinion of the Principal Investigator, may cause undue risk to the subject
10. Other: Any condition or characteristic that in the judgment of the Principal Investigator would create a logistical or safety contraindication to enrollment (e.g., shoulder width greater than the bore of the MRI or PET/MRI machines)

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males, regardless of race or ethnicity, currently serving in the Special Operation Forces
Study Population: U.S. Special Operations Forces personnel
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Diffusion MRI structural connectivity | Day 1
  measured by white matter tractography
fMRI resting state functional connectivity | Day 2
  measured by default mode network connectivity
PET Neuroinflammation | Day 1
  measured by standardized uptake value ratio of TSPO ligand [11C]PBR28
PET Tau deposition | Day 2
  measured by standardized uptake value ratio of [18F]MK6240
Neurofilament Light Chain | Day 1, after 6-8 hour fasting
  measured by serum concentration of neurofilament light chain
Cognitive Function | Day 1
  measured by the Trail Making Test
Behavioral symptoms | Day 2
  measured by the Neurobehavioral Symptom Inventory
Physical symptoms | Day 2
  measured by the Neurobehavioral Symptom Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Edlow, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States